CLINICAL TRIAL: NCT05923892
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Trial to Evaluate the Efficacy and Safety of Different Doses of OPS-2071 in the Treatment of Irritable Bowel Syndrome of Diarrhea Type (IBS-D)
Brief Title: Phase II Clinical Trial of OPS-2071 in the Treatment of Irritable Bowel Syndrome of Diarrhea Type
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 341-403-00010
Record Dates: First submitted 2023-01-11; First posted 2023-06-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-04

CONDITIONS: Irritable Bowel Syndrome of Diarrhea Type (IBS-D)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3 dose groups of OPS-2071 (Experimental): OPS-2071 tablets, 50 mg OPS-2071 tablets, 100 mg OPS-2071 tablets, 200 mg Take 4 tablets/bid, after meals in the morning and evening, with an interval of at least 8 hours for 2 weeks(The dosing interval will be 12 hours from Day 5 to Day 7).
  Interventions: Drug: OPS-2071
- placebo group (Placebo Comparator): Placebo tablets Take 4 tablets/bid, after meals in the morning and evening, with an interval of at least 8 hours for 2 weeks(The dosing interval will be 12 hours from Day 5 to Day 7).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: OPS-2071 — There are 3 dose groups of OPS-2071，OPS-2071 tablets, 50 mg、100mg、200mg. Take 4 tablets/bid, after meals in the morning and evening, with an interval of at least 8 hours for 2 weeks(The dosing interval will be 12 hours from Day 5 to Day 7).
  Other Names: OPS-2071 tablets
  Arms: 3 dose groups of OPS-2071
Drug: placebo — Take 4 tablets/bid, after meals in the morning and evening, with an interval of at least 8 hours for 2 weeks(The dosing interval will be 12 hours from Day 5 to Day 7).
  Other Names: placebo tablets
  Arms: placebo group

SUMMARY:
This is a A Multicenter, Randomized, Double-blind, Placebo-controlled, Clinical Trial to Evaluate the Efficacy and Safety of Different Doses of OPS-2071 in the Treatment of Irritable Bowel Syndrome of Diarrhea type (IBS-D).The trial is mainly divided into three periods: screening period, treatment period and follow-up period.

DETAILED DESCRIPTION:
Screening period:

After signing the Informed Consent Form, subjects entered a 14-day screening period to evaluate inclusion/exclusion criteria and collect demographic information, medical history, etc. Subject's previous medication should be eluted and concomitant medications should be prohibited.

Treatment period:

After the screening period, subjects who meet the inclusion criteria and do not meet the exclusion criteria will be randomly assigned (1:1:1:1) to four treatment groups to receive a 2-week treatment period. Weekly follow-up and relevant examinations will be performed.

Follow-up period:

The safety follow-up visit will be conducted by telephone on Day14 (+2) after the last dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able to fully understand and willing to comply with the trial procedures, and voluntarily participate in the trial and sign the Informed Consent Form;
2. Subjects aged 18 to 65 years at the time of ICF signing;
3. Subjects who meet Rome IV diagnostic criteria for IBS-D;
4. The following criteria should be met during the screening period:

Exclusion Criteria:

1. Subjects who have gastrointestinal alarm symptoms within 14 days before screening, such as hematochezia, positive fecal occult blood test, anemia, abdominal mass, ascites, fever, unexplained body mass loss, and nocturnal diarrhea;
2. Subjects with previously confirmed diagnosis of digestive organic diseases, such as inflammatory bowel disease, intestinal tuberculosis, intestinal polyps (except for polyps ≤ 0. 3 cm or polypectomy time ≥ 15 days), intestinal diverticulum, intestinal tumor, etc., or patients still complicated with peptic ulcer and infectious diarrhea;
3. Subjects with previously confirmed diagnosis of diseases affecting digestive system function, such as uncontrolled hyperthyroidism or hypothyroidism, chronic renal failure, autoimmune diseases, diabetes, and neurological (such as anorexia nervosa) or serious psychiatric system diseases (such as major depression or severe anxiety);
4. Subjects with previously confirmed diagnosis of diseases with symptoms similar to IBS, such as eosinophilic enteritis, microscopic colitis (including collagenous colitis and lymphocytic colitis), lactose intolerance, malabsorption syndrome, etc.;
5. Subjects with previously confirmed diagnosis of non-intestinal digestive diseases, such as tuberculous peritonitis, gallstones, cirrhosis, chronic pancreatitis, etc.;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 2 in NRS (Numerical rating scale,0-10 points,higher scores mean a worse outcome )abdominal pain. | 2 week
  Efficacy is defined as ≥ 30% improvement in abdominal pain symptoms compared to baseline.
Change from baseline to Week 2 in Bristol（type 1 to type 7，higher type means worse）stool scale. | 2 week
  Efficacy is defined as ≥ 50% reduction in the number of days with at least one stool that has a consistency of Bristol stool scale of 6 or 7 for at least 50% of the treatment period.

SECONDARY OUTCOMES:
Improvement degree of abdominal pain and abnormal defecation (%) | 2 week
  abdominal pain (0-100%,higher degree means better) and abnormal defecation (0-100%,0-100%,higher degree means better)
Abdominal pain score and days of abdominal pain remission | 2 week
  will be collected from Record of severity of IBS symptoms which included the severity of abdominal pain(from 0 to 100%,higher degree means worse) and the day of abdominal pain in the past 10 days
Changes in defecation frequency | 2 week
  will be collected from Record of defecation frequency
Changes in and abdominal distension | 2 week
  will be collected from Record of severity of IBS symptoms which included abdominal distension(0-10, higher degree means worse)
Subject's subjective response | 2 week
  will be collected from Record of severity of IBS symptoms which included the subject's satisfacation degree of his defecation habbit(0-100%) and the influence of the IBS symptoms in his life(0-100%)
Detection of intestinal flora | 2 week
  Macrogenomic detection to detect the change of intestinal flora
defecation urgency | 2 week
  will be collected from Record of severity of IBS symptoms which included the defecation urgency(0-10) of the past 10 days
fecal property | 2 week
  will be collected from Record of bristol scale( from type1 to type7, higher type means worese)

CONTACTS AND LOCATIONS:
Overall Officials: Hou xiaohua, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No